CLINICAL TRIAL: NCT05230121
Title: Intestinal Dysmotility in Patients With Functional Digestive Symptoms: Significance of Minute Rythm
Brief Title: Intestinal Dysmotility: Minute Rythm
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: PR(AG)56/2018D
Record Dates: First submitted 2022-01-11; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Motility Disorder of Small Intestine (Disorder)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Intestinal manometry may detect phasic pressure patterns that suggest small bowel obstruction. The most common is the "clustered contractions pattern", characterized by repetitive short spouts of intestinal contractions in the postprandial period. When encountered in patients with chronic unexplained digestive symptoms, an exhaustive radiological evaluation of the gut should be performed to exclude partial mechanical obstruction. If no luminal compromise is identified by the imaging studies, an underlying neuropathic disorder of the bowel may be the probable diagnosis. The objective of this study was to determine the clinical significance of this pattern in patients evaluated for a possible intestinal motility disorder. Study design: Retrospective analysis of the of patients with minute rhythm pattern detected in intestinal manometric recordings performed between 2010 and 2018 at the Vall d'Hebron Digestive Function Unit in consecutive patients referred for evaluation of intestinal motility due to severe, chronic digestive symptoms and suspected dysmotility. The manometric recordings that had been informed of minute rhythm pattern, will be retrieved to confirm the original report. The clinical records of these patients will be reviewed to obtain: a) demographic data, b) digestive symptoms at the time of evaluation, c) history of abdomino-pelvic surgeries or radiotherapy prior to manometry, d) diagnosis of systemic disorders, and e) presence of esophageal, gastric or colonic dysmotility. Results from radiological and other investigations will be also revised, as well as therapeutic decisions and clinical outcome. Particularly, whether abdominal imaging studies (simple abdominal X-ray or abdominal CT scans) were performed within 7 days of the manometric study, and whether these studies showed signs of fecal retention (presence of solid stools in the right colon) or not.

ELIGIBILITY:
Inclusion criteria:

- Patients with minute rhythm pattern by intestinal manometry, defined as short clusters of 3-5 contractions repeating every 1-3 min and occurring over a ≥ 20-cm intestinal segment during a ≥ 30-min period in postprandial conditions.

Exclusion criteria:

* Patients with an incomplete (< 2 hour) postprandial recording.
* Patients with minute rhythm detected exclusively in fasting conditions or lasting less than 30 min in postprandial conditions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with minute rhythm pattern detected in intestinal manometric recordings performed between 2010 and 2018 at the Vall d'Hebron Digestive Function Unit in consecutive patients referred for evaluation of intestinal motility due to severe, chronic digestive symptoms and suspected dysmotility.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
fecal retention | 7 days
  Presence of solid stools in the right colon in abdominal imaging studies (simple abdominal X-ray or abdominal CT scans) performed within 7 days of the manometric study

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No